CLINICAL TRIAL: NCT03785535
Title: Functional MRI Study of the Effects of Vibrotactile Sensory Stimulation on Brain Activity in Fibromyalgia Patients
Brief Title: Functional MRI Study of Vibrotactile Stimulation Effects in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovoxel SLP (Other)
Responsible Party: Principal Investigator, Jesus Pujol, Principal Investigator, Neurovoxel SLP
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSI2017-83777-P
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual treatment (Experimental): Vibrotactile sensory stimulation will consist on whole-body stimulation with mechanical stimuli of pallesthetic type at high rate (2-90 Hz), low intensity and long daily duration (3h).
  Interventions: Device: Vibrotactile stimulation
- Sham (Sham Comparator): Sham treatment will be applied using identical instruments and with power and duration programmed identically. However, in this case, the output will not be the signal activating the vibration motors, but rather an electrical signal turning on an incorporated pilot light indicating that the (simulated) treatment was operating
  Interventions: Device: Vibrotactile stimulation

INTERVENTIONS:
Device: Vibrotactile stimulation — The active treatment will involve whole-body sensory stimulation with mechanical stimuli of vibrotactile (pallesthetic) type at a relatively high rate, low intensity and long duration administered at sleep time (a total daily duration of 3 h distributed within a period of 2 h at bedtime and 1 h prior to getting up). The intensity will be 30% of power at bedtime and 45% prior to getting up.

SUMMARY:
The purpose of this study is to investigate the effects of low-intensity and prolonged vibrotactile sensory stimulation on brain activity and functional connectivity in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of fibromyalgia according to the American College of Rheumatology (ACR) (Arthritis Care Res 2010;62:600-10).
2. Clinical symptoms are not a consequence of other medical disorder (although the presence of other disorders is not an exclusion criterion)
3. Diagnoses established by an expert on fibromyalgia.
4. Stable treatment of chronic use.
5. Subject demonstrates an understanding of the study and a willingness to participate as evidenced by voluntary written informed consent.

Exclusion Criteria:

1. Generalized inflammatory articular or rheumatic disease.
2. Severe, non-stable medical, endocrinological or neurological disorder.
3. Psychotic disorder or drug abuse.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Functional MRI measures of brain functional connectivity. A correlation scale ranging from 0 to 1 will be used. | 3 weeks
  Change on brain activity rated using functional MRI measures of functional connectivity
Functional MRI measures of brain activity. A functional MRI signal change scale ranging from 0 to 1 will be used. | 3 weeks
  Change on brain activity rated using functional MRI measures of brain activation in response to nociceptive stimulation

SECONDARY OUTCOMES:
Functional MRI measures of sensory system activity. A functional MRI signal change scale ranging from 0 to 1 will be used. | 3 weeks
  Change on brain activity rated using functional MRI measures of brain activation in response to non-nociceptive stimulation
Measured fibromyalgia symptoms using a 101-point numerical rating scale. | 3 weeks
  Change on fibromyalgia symptoms (including pain, fatigue, cognitive symptoms, sleep disturbance, and general health rating). Rated using Numerical Rating 101-point Scales.
Tolerability rated using a numerical rating scale ranging from 0 to 100 points. | 3 weeks
  Tolerability index (0-100).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain